CLINICAL TRIAL: NCT05999253
Title: Comparison of the Effects of Modified Thoracolumbar Interfacial Plane (mTLIP) Block and Erector Spina Plane Block on Postoperative Pain and Opioid Analgesic Consumption in Patients Undergoing Lumbar Discectomy for Lumbar Disc Herniation
Brief Title: Comparison of the Efficacy of Thoracolumbar Interfascial Plane Block and Erector Spina Plane Block in Lumbar Discectomy
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil, Anesthesiology and Reanimation Spesialist, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 05.05.2023/373
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified thoracolumbar plane block (mTLIP): Modified thoracolumbar plane block (mTLIP): under ultrasound-guided, the lateral compartment of the longissimus muscle and iliocostal muscle muscles are imagined and the block needle is placed in the interfascial plane of these two muscles and local anesthesic solution is appliced.
  * Patients will be induced with standard general anesthesia and turned to the prone position.
  * Before the surgical incision, 20 ml of 0.25% bupivacaine 0.25% will be administered bilaterally under ultrasound guidance only once.
  * 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
  * Plane block applications will be performed by anaesthesiologists with at least 5 years of experience
  Interventions: Procedure: Modified thoracolumbar plane block (mTLIP)
- Erector spinae plane block (ESP): Erector spinae plane block (ESP): After determining the vertebral spinal process and trapezius, rhomboid major and erector spinae muscles with ultrasound guidance, the block needle is advanced in the cranio-caudal direction with an in plane approach and local anaesthetic solution is applied to the plane between the erector spinae muscle and the transverse process when the needle rests on the transverse process.
  * Patients will be induced with standard general anesthesia and turned to the prone position.
  * Before the surgical incision, 20 ml of 0.25% bupivacaine will be administered bilaterally under ultrasound guidance only once.
  * 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
  * Plane block applications will be performed by anaesthesiologists with at least 5 years of experience
  Interventions: Procedure: Erector spinae plane block (ESP)

INTERVENTIONS:
Procedure: Modified thoracolumbar plane block (mTLIP) — Modified thoracolumbar plane block (mTLIP): under ultrasound-guided, the lateral compartment of the longissimus muscle and iliocostal muscle muscles are imagined and the block needle is placed in the interfascial plane of these two muscles and local anesthesic solution is appliced.
  * 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
  * to be administered only approximately 20-30 minutes before the onset of anaesthesia.
  Other Names: Plane block
  Groups: Modified thoracolumbar plane block (mTLIP)
Procedure: Erector spinae plane block (ESP) — Erector spinae plane block (ESP): After determining the vertebral spinal process and trapezius, rhomboid major and erector spinae muscles with ultrasound guidance, the block needle is advanced in the cranio-caudal direction with an in plane approach and local anaesthetic solution is applied to the plane between the erector spinae muscle and the transverse process when the needle rests on the transverse process.
  * 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
  * to be administered only approximately 20-30 minutes before the onset of anaesthesia
  Other Names: Plane block
  Groups: Erector spinae plane block (ESP)

SUMMARY:
Patients who will undergo herniated disc surgery have serious pain after surgery. In order to minimise this pain and to ensure that they recover more quickly and use less morphine-derived painkillers, we aim to apply two types of painkiller injections before surgery. For this purpose, it is planned to apply painkiller injections on both sides of the level of the herniated disc with sedation before the operation. Afterwards, herniated disc surgery will be performed under general anaesthesia.

DETAILED DESCRIPTION:
Modified thoracolumbar plane block (mTLIP): under ultrasound-guided, the lateral compartment of the longissimus muscle and iliocostal muscle muscles are imagined and the block needle is placed in the interfascial plane of these two muscles and local anesthesic solution is appliced.

* 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
* to be administered only approximately 20-30 minutes before the onset of anaesthesia.
* only once in the preoperative block room approximately 20-30 minutes before induction of anaesthesia
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* patients' intraoperative fentanyl consumption, agitation-sedation scores on awakening from anaesthesia, tramadol consumption in the postoperative 24 hours, postoperative VAS pain scores, and side effects such as postoperative nausea-vomiting will be evaluated.
* plane blocks will be applied under ultrasound guidance.
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* Postoperative evaluations of patients will be performed face to face. Patients will be routinely administered 1 g paracetamol intravenously at 8 hour intervals in the postoperative period. 100 mg tramadol intravenously will be administered if their pain is above VAS 4 despite this.
* This study was followed up in the neurosurgery unit of SBU Gazi Yasargil Training and Research Hospital.
* Patients were sedated with 1 mg midazolam and 50 mcg fentanyl intravenously in the preoperative preparation room in the operating room and 20 ml of 0.25% bupivacaine was administered bilaterally on each side under ultrasound guidance. After the block application, the patient was taken to the operating room and standard general anaesthesia was applied.

Patients will be monitored for pain and side effects at the neurosurgery unit , 1st hour, 2nd hour, 4th hour, 8th hour and 24th hour in the postoperative period.

- Both plan blocks are applied for analgesia in the postoperative period and aim to reduce opioid consumption in the postoperative period.

Erector spinae plane block (ESP): After determining the vertebral spinal process and trapezius, rhomboid major and erector spinae muscles with ultrasound guidance, the block needle is advanced in the cranio-caudal direction with an in plane approach and local anaesthetic solution is applied to the plane between the erector spinae muscle and the transverse process when the needle rests on the transverse process.

* 20 ml of 0.25% bupivacaine will be used on each side (total of 40 ml of 0.25% bupivacaine will be used)
* to be administered only approximately 20-30 minutes before the onset of anaesthesia.
* only once in the preoperative block room approximately 20-30 minutes before induction of anaesthesia
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* patients' intraoperative fentanyl consumption, agitation-sedation scores on awakening from anaesthesia, tramadol consumption in the postoperative 24 hours, postoperative VAS pain scores, and side effects such as postoperative nausea-vomiting will be evaluated.
* plane blocks will be applied under ultrasound guidance.
* plane block applications will be performed by anaesthesiologists with at least 5 years of experience
* Postoperative evaluations of patients will be performed face to face.

Statistical methods / analysis: G-Power version 3.1.9.4 (Universität Kiel, Germany) program was used to calculate the sample size. The two-tailed alpha error was taken as 0.05, power as 0.80 and effect size as 0.8, and based on a previous study the allocation ratio was accepted as N2/N1:1. The minimum number of patients to be included in the study was calculated as 72.

SPSS 16.0 for Windows (SPSS Inc., Chicago, IL, USA) was used for other statistical analyses. Statistical data were expressed as mean and standard deviation, while categorical data were expressed as frequency and percentage. Comparison of categorical data in the groups was done with Chi-square, the results were given as %n. Shapiro-Wilk tests were used to determine if the numerical data fit the normal distribution. While the data fitting the normal distribution were evaluated with the Student's t-test. Mann- Whitney U tests were used to compare the data differ from the normal distribution. p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years of age, ASA I-III, scheduled for Lumbar Disc Herniation operation under general anaesthesia.

Exclusion Criteria:

* ASA >III body mass index (BMI) > 35 kg/m2 known allergy to local anaesthetics presence of preoperative chronic pain presence of coagulopathy those who are unable to give written consent non-voluntary patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be operated for 1 or 2 level lumbar disc herniation.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | assessed at postoperative 1st, 2nd, 4th, 8th and 24th hours
  * The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
  * Low back pain and leg pain as an extension of the traveling nerve assessed using visual pain scores (VAS) will be evaluated

SECONDARY OUTCOMES:
Sedation- agitation level | After extubation]
  The Riker Sedation- Agitation Scale (RSAS): identifies seven levels of sedation and agitation, which range from dangerous agitation to deep sedation, with a thorough description of patient behavior.
  Riker sedation-agitation Scale:1- Unarousable, 2 -Very Sedated, 3- Sedated, 4 Calm and Cooperative, 5 -Agitated, 6 -Very Agitated, 7 -Dangerous Agitation
Nausea-vomiting | postoperative 1st, 2nd, 4th, 8th and 24th hours
  -Postoperative nausea and vomiting will be assessed using a 100 mm Visual Analogue Scale (VAS):
  1- severe nausea (VAS>70 mm), 2- moderate nausea (50<VAS<70 mm), 3- mild nausea (VAS <50 mm).
Systolic, diastolic and mean arterial pressure monitoring | before the start of surgery, at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes, 40 minutes, 50th minutes, 60 minutes after the start of surgery
  Blood pressure will be measured with a non-invasive automatic pneumatic cuff in the operating theatre.
heart rate monitoring | before the start of surgery, at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes, 40 minutes, 50th minutes, 60 minutes after the start of surgery
  the measurement will be obtained by electrocardiographic monitoring
amount of fentanyl consumed during the operation | during surgery
  micrograms of fentanyl consumed
Amount of tramadol used postoperatively | during the postoperative 24 hour]
  Amount of tramadol used postoperatively (milligrams)
Surgery duration | at the end of surgery]
  Time in hours from the start of the surgical incision until the last surgical suture is placed
Anesthesia duration | at the end of anaesthesia]
  time in hours from induction of anaesthesia to extubation
patient satisfaction assessmen | at the end of 24 hours postoperatively
  Patients' satisfaction with the quality of pain management will be assessed at 24 hours postoperatively using the following scale:
  1 = very dissatisfied; 2 = quite dissatisfied; 3 = moderate; 4 = quite satisfied; 5 = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Cem K. Kaçar, Assoc.Prof, Study Director — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
* after de-identification; all individual participant data collected during the research and the primary and secondary outcomes of the study.
  * data can be shared immediately after publication, no end date set.
  * case-by-case basis at the discretion of Primary Sponsor
  * data can be access subject to approvals by Principal Investigator (e-mail: fatma.acil@saglik.gov.tr)

REFERENCES:
- [Background] Ciftci B, Ekinci M, Celik EC, Yayik AM, Aydin ME, Ahiskalioglu A. Ultrasound-Guided Erector Spinae Plane Block versus Modified-Thoracolumbar Interfascial Plane Block for Lumbar Discectomy Surgery: A Randomized, Controlled Study. World Neurosurg. 2020 Dec;144:e849-e855. doi: 10.1016/j.wneu.2020.09.077. Epub 2020 Sep 18. PMID 32956890